CLINICAL TRIAL: NCT04254770
Title: A Randomized, Parallel-design Study to Evaluate the Effects of Home Use of the Sonicare Powered Toothbrush and a Manual Toothbrush on Subjects With Periodontitis
Brief Title: At-Home Care for Subjects With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OHC_OHC_Anthony_2019_10606
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Periodontitis; Dental Plaque
MeSH Terms: conditions — Periodontitis; Dental Plaque

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADA (American Dental Association) approved Manual Toothbrush (Active Comparator)
  Interventions: Device: ADA approved Manual Toothbrush
- Marketed Power Toothbrush (Experimental)
  Interventions: Device: Marketed Power Toothbrush

INTERVENTIONS:
Device: ADA approved Manual Toothbrush — ADA approved Manual Toothbrush
  Arms: ADA (American Dental Association) approved Manual Toothbrush
Device: Marketed Power Toothbrush — Marketed Power Toothbrush
  Arms: Marketed Power Toothbrush

SUMMARY:
The effect of use of powered toothbrushing in patients exhibiting periodontal inflammation has been observed repeatedly in clinical studies conducted over a 20+ year period. Whether these subjects also had periodontitis, or not, was not a collected data metric as it was outside the scope of the Investigation. This study, therefore, will specifically include and document that a subject exhibits periodontitis upon study entry, and measure the ensuing response following professional treatment of scaling and root planing, followed by home use of the assigned study products (powered or manual toothbrushing).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-75 years
* Exhibiting Stage I or II periodontitis
* Minimum of 20 'scorable' teeth (excluding 3rd molars)
* Regular manual toothbrush user
* Have a minimum average plaque score of > 1.8 per Modified Plaque Index scoring with 3-6 hours plaque accumulation
* Agree to desist use of interproximal cleaning aids and other prohibited devices or medicaments during the study period
* Be a non-smoker (> 10 years), or never smoker

Exclusion Criteria:

* Have a cardiac pacemaker or implanted cardiac defibrillator
* Have uncontrolled Insulin-Dependent Diabetes Have current use of antibiotic medications or use within 4 weeks of enrollment
* Have current use of prescription-dose anti-inflammatory medications or anticoagulants Have excessive gingival recession, per Investigator/Examiner discretion
* Have heavy deposits of calculus, either supragingival and/or subgingival, per Investigator/Examiner discretion
* Have had a professional prophylaxis within 4 weeks of the study
* Prior chemotherapy, immunotherapy or radiation therapy within last 10 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Change in symptoms of inflammation of the periodontium, as measured by Bleeding on Probing. | 6 months

SECONDARY OUTCOMES:
Change in supragingival plaque, as measured by Modified Plaque Index | 6 months
Change in clinical attachment level | 6 months
Change in periodontitis, as measured by probing pocket depth | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Inc, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jenkins W, Starke EM, Nelson M, Milleman K, Milleman J, Ward M. The effects of scaling and root planing plus home oral hygiene maintenance in Stage I/II periodontitis population: A 24-week randomized clinical trial. Int J Dent Hyg. 2024 Aug;22(3):727-735. doi: 10.1111/idh.12783. Epub 2024 Jan 30. PMID 38289823